CLINICAL TRIAL: NCT04547855
Title: A Phase II Study of Anlotinib Combined With Dose-dense Temozolomide for the First Recurrent or Progressive Glioblastoma After STUPP Regimen
Brief Title: Anlotinib Combined With Dose-dense Temozolomide for the First Recurrent or Progressive Glioblastoma After STUPP Regimen
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonggao Mou (Other)
Collaborators: The First Affiliated Hospital of Nanchang University (Other)
Responsible Party: Sponsor-Investigator, Yonggao Mou, MD, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Qun-Ying YANG
Record Dates: First submitted 2020-09-11; First posted 2020-09-14 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental group (Experimental): anlotinib combined with dose-dense temozolomide
  Interventions: Drug: anlotinib combined with dose-dense temozolomide

INTERVENTIONS:
Drug: anlotinib combined with dose-dense temozolomide — Temozolomide Capsule 150mg, p.o., qd, d1-7,15-21,4 weeks one cycle; Anlotinib hydrochloride capsule 12mg, p.o., qd, D1-D14; 3 weeks one cycle.
  Other Names: Anlotinib hydrochloride capsule

SUMMARY:
Currently,6 cycles of Temozolomide adjuvant chemotherapy after concurrent radiotherapy and Temozolomide chemotherapy(STUPP regimen)for newly diagnosed postoperative GBM can increase the 2-year and 5-year overall survival rates of patients to 26.5% and 9.8%, respectively. However, most patients are still unable to avoid tumor recurrence and death.Anlotinib is an efficient multi-target tyrosine kinase inhibitor (TKI) that effectively block the migration and proliferation of endothelial cells and reduce tumor microvascular density by targeting VEGFRs, FGFRs, PDGFRs. It has been proved to be safe and effective in advanced lung cancer(including NSCLC,SCLC)after second-line standard chemotherapy failure,and advanced soft tissue sarcoma after anthracycline-containing chemotherapy failure.Here, we prepared to evaluate whether the combination of dose-dense Temozolomide and Anlotinib can preferably improved survival of the first recurrent or progressive GBM after STUPP regimen.

ELIGIBILITY:
Inclusion Criteria:

1. The primary tumor must be pathologically confirmed as supratentorial glioblastoma;
2. The primary tumor progressed or relapsed for the first time after surgery (including biopsy, partial resection, total resection), standard radiotherapy and temozolomide concurrent chemotherapy and temozolomide adjuvant chemotherapy (STUPP regimen), including multiple intracranial recurrence and new lesions.;
3. Age ≥ 18 years old,≤75 years old;
4. KPS ≥ 60;
5. the expected survival time is more than 12 weeks;
6. within 28 days before entering the group, patients need to undergo craniocerebral enhanced MRI, and the lesions on MRI must be measurable;
7. for patients undergoing the second surgery after the first recurrence, baseline MRI should be obtained at least 4 weeks after operation;
8. if the patient is undergoing hormone therapy, the hormone dose must be stable or reduced at least 5 days before baseline MRI;
9. For patients undergoing re-radiation therapy, the baseline MRI should be obtained at least 8 weeks or 4 weeks after the end of the radiotherapy (the recurrence lesion is not in the radiation field);
10. For patients who are treated with gamma knife or other hyperdivision methods for the first time, Recurrence or progression must be confirmed by pathology (except for patients with new lesions);
11. Peripheral blood picture, liver and kidney function, etc. are within the following allowable range (detected within 7 days before the start of treatment): neutrophils (ANC) ≥ 1.5×109/L; hemoglobin (HGB) ≥100g/L; platelets (PLT) ≥100×109/L; liver transaminase (AST/ALT) ≤2.5 times the upper limit of the normal range; total bilirubin (TBIL) <1.5 times the upper limit of the normal range; Creatinine (CREAT) <1.2 times the upper limit of the normal range; International normalized ratio (INR) <1.5; Activated partial thromboplastin time (APTT) <1.5 times the upper limit of the normal range (except for patients receiving anticoagulation therapy); Urinary protein (PRO)/creatinine (CRE) ratio ≤1.0;
12. The patient must have fully recovered from the toxicity of previous chemotherapy or targeted therapy, and at least 30 days from the last treatment; 13.Before starting treatment, the patient must Complete recovery from surgery, postoperative infection or other comorbidities;

14.Patients of childbearing age (including female and male patients' female partners) must take effective birth control measures; 15.Sign informed consent.

Exclusion Criteria:

* 1.Patients who have participated in other clinical trials in the past and have not terminated the trial; 2.Patients who have used Anlotinib in the past; 3. Baseline MRI suggests the recent risk of cerebral hemorrhage or brain herniation; 4. Pregnant or breast-feeding women; 5.Those who are difficult to control acute infections; 6. People who take drugs, drug abuse, long-term alcoholism and AIDS; 7.Have frequent vomiting or have conditions that affect the oral administration of drugs; 8. Hypertension that cannot be controlled by drugs The patient (>150/100mmHg); 9. Previous hypertensive encephalopathy; 10. Hemorrhage tendency or coagulopathy; 11. Thrombolytic or anticoagulant therapy (unless low molecular weight heparin or warfarin is used); 12).≥ Grade 2 cardiac insufficiency (NYHA criteria) or congestive heart failure; 13. Past history of myocardial infarction or unstable angina, stroke and transient ischemic attack within 6 months; 14. Serious vascular disease; 15.Peripheral artery embolism occurred recently; 16. Abdominal fistula, gastrointestinal perforation and abdominal abscess occurred in the past; 17.Intracranial abscess occurred within 6 months; 18. Major surgery, open biopsy or Have suffered major trauma; 19. Those who are expected to undergo major surgery; 20).Those who have severe incurable wounds, ulcers or fractures; 21).Those with a history of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonia, drug-related pneumonia, severely impaired lung function, etc.; 22.patients who are allergic to known ingredients of Anlotinib; 23.There is a serious skin disease; 24. Other concomitant diseases that seriously endanger the safety of patients or affect the completion of the study according to the judgment of the investigator .

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2020-09-11 (Actual); Primary Completion 2022-09-11 (Estimated); Study Completion 2023-03-11 (Estimated)

PRIMARY OUTCOMES:
6 months Objective Response Rates | 6 month
  Percentage of Participants With Objective Response (Partial Response [PR] Plus Complete Response [CR]), as Assessed Using as Assessed by Investigator Using RANO Version 1.1
6 months Progression-Free Survival Rates | 6 months
  6 months Progression-Free Survival Rates as Assessed by Investigator Using RANO Version 1.1

SECONDARY OUTCOMES:
Progress-free survival (PFS) | Approximately 6 months
  Progression-Free Survival (PFS) as Assessed by Investigator Using RANO Version 1.1
overall survival | Approximately 1 years
  OS was defined as the time from the date of randomization to the date of death due to any cause.
Toxic side effects | Approximately 1 years
  Toxic side effects as Assessed by Investigator Using RANO Version 1.1

CONTACTS AND LOCATIONS:
Overall Officials: QUN-YING YANG, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: 1 year